CLINICAL TRIAL: NCT07203794
Title: A Prospective, Randomized Controlled Study Comparing the Analgesic Efficacy of Bupivacaine Infiltration of the Gallbladder Bed and Trocar Sites, Erector Spinae Plane Block, and Intrathecal Morphine in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Analgesic Efficacy of Bupivacaine Infiltration, Erector Spinae Plane Block, and Intrathecal Morphine in Laparoscopic Cholecystectomy
Acronym: ITM-ESP-IPLA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, irem ateş, Associate Professor as the Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/616; 2025/2 (Other: Atatürk University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-09-22; First posted 2025-10-02 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain Management; Cholecystectomy, Laparoscopic
Keywords: Laparoscopic Cholecystectomy; Postoperative Pain; Bupivacaine Infiltration; Erector Spinae Plane Block; Intrathecal Morphine; Analgesia; Opioid Consumption
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine; Anesthesia, Conduction

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized, parallel-group, controlled trial with three intervention arms. Eligible patients undergoing elective laparoscopic cholecystectomy will be randomly assigned in a 1:1:1 ratio to receive either bupivacaine infiltration of the gallbladder bed and trocar sites, bilateral ultrasound-guided erector spinae plane block, or intrathecal morphine. Each participant will receive only one of the three interventions in addition to standard general anesthesia and multimodal analgesia. The outcomes will be compared across groups to evaluate the relative analgesic efficacy of the interventions.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and postoperative outcome assessors will be blinded to group allocation. The anesthesiologist performing the intervention cannot be blinded due to the nature of the procedures, but will not be involved in postoperative data collection or outcome assessment. Thus, the trial will be conducted with patient- and assessor-blinding to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bupivacaine Infiltration Group (Active Comparator): Patients will receive bupivacaine infiltration at the gallbladder bed and trocar sites following laparoscopic cholecystectomy. After removal of the gallbladder, 20 mL of 0.25% bupivacaine will be applied to the gallbladder bed using a sterile sponge for 10-15 minutes. At the end of surgery, a total of 20 mL 0.25% bupivacaine will be infiltrated at trocar insertion sites (8 mL umbilical port, 6 mL epigastric port, 3 mL each auxiliary port).
  Interventions: Drug: Bupivacaine Infiltration
- Erector Spinae Plane Block Group (Active Comparator): Patients will undergo bilateral erector spinae plane block under ultrasound guidance before induction of anesthesia. Under ultrasound guidance at the T7 transverse process level, a total of 40 mL of 0.25% bupivacaine will be injected bilaterally using an in-plane technique prior to induction of anesthesia.
  Interventions: Procedure: Erector Spinae Plane Block
- Intrathecal Morphine Group (Active Comparator): Patients will receive intrathecal morphine prior to induction of anesthesia. With the patient in a sitting position, a 27G spinal needle will be inserted at the L3-L4 interspace, and 200 mcg of morphine will be administered intrathecally before induction of anesthesia.
  Interventions: Drug: Intrathecal Morphine

INTERVENTIONS:
Drug: Bupivacaine Infiltration — After removal of the gallbladder, 40 mL of 0.25% bupivacaine will be applied to the gallbladder bed with a sterile sponge for 10-15 minutes. At the end of the surgery, 15 mL of 0.25% bupivacaine will be infiltrated into trocar insertion sites (5 mL umbilical port, 5 mL epigastric port, 5 mL each auxiliary port).
  Other Names: Marcaine; Local Infiltration
  Arms: Bupivacaine Infiltration Group
Procedure: Erector Spinae Plane Block — Before induction of anesthesia, a bilateral ultrasound-guided erector spinae plane block will be performed at the T7 transverse process level. A total of 40 mL of 0.25% bupivacaine will be injected (20 mL per side) using an in-plane technique under ultrasound guidance.
  Other Names: ESP Block; Regional Anesthesia
  Arms: Erector Spinae Plane Block Group
Drug: Intrathecal Morphine — With the patient in the sitting position, a 27-gauge spinal needle will be inserted at the L3-L4 interspace. A dose of 100 mcg morphine will be administered intrathecally before induction of anesthesia.
  Arms: Intrathecal Morphine Group

SUMMARY:
This study is designed to compare three different methods of pain control after laparoscopic gallbladder surgery (laparoscopic cholecystectomy). Although this surgery is minimally invasive, participants often experience different types of pain after the operation, such as pain at the incision site, pain inside the abdomen, and shoulder pain caused by the gas used during surgery.

The investigators will compare three commonly used pain relief techniques:

Local infiltration - injecting a numbing medicine (bupivacaine) into the gallbladder bed and at the sites where the surgical instruments are placed.

Erector spinae plane (ESP) block - an ultrasound-guided nerve block performed in the back to reduce both abdominal and incisional pain.

Intrathecal morphine - a very small dose of morphine given into the spinal fluid before surgery to provide long-lasting pain relief.

The goal is to determine which method provides the best pain control, reduces the need for opioid medications, and improves recovery after surgery.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is the standard surgical treatment for gallbladder diseases. Despite being a minimally invasive procedure, postoperative pain is a frequent problem and can negatively affect early mobilization, oral intake, and overall recovery. The pain experienced after this surgery is multifactorial, including somatic pain at trocar sites, visceral pain at the gallbladder bed, and shoulder pain caused by carbon dioxide insufflation. Effective pain management is therefore essential to improve patient comfort, reduce opioid consumption, and shorten hospital stay.

Several methods are available for postoperative analgesia. Local infiltration of the gallbladder bed and trocar sites with bupivacaine provides targeted pain relief at areas of surgical trauma. Erector spinae plane (ESP) block, a recently described ultrasound-guided regional anesthesia technique, offers both somatic and visceral analgesia with a favorable safety profile. Low-dose intrathecal morphine has also been shown to provide strong and prolonged analgesia in abdominal surgery, though its use may be limited by side effects such as nausea, vomiting, and itching.

This single-center, prospective, randomized controlled trial will compare the analgesic efficacy of three techniques:

Group INF (Infiltration): Bupivacaine infiltration at the gallbladder bed and trocar sites.

Group ESP: Bilateral ultrasound-guided ESP block at the T7 level.

Group ITM: Intrathecal morphine administration before induction of anesthesia.

The primary outcome is total opioid consumption within the first 24 hours after surgery.

Secondary outcomes include postoperative pain scores at multiple time points using the Visual Analog Scale (VAS), as well as the incidence of side effects such as nausea, vomiting, pruritus, and respiratory depression.

The results of this study are expected to provide evidence to guide multimodal analgesia strategies in laparoscopic cholecystectomy and to optimize patient recovery and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Scheduled for elective laparoscopic cholecystectomy
* American Society of Anesthesiologists (ASA) physical status I-III
* Able to provide written informed consent

Exclusion Criteria:

* Body mass index (BMI) > 35 kg/m²
* History of coagulopathy or bleeding disorders
* Known allergy or hypersensitivity to opioids or local anesthetics
* Chronic pain or regular analgesic use
* History of neurological or psychiatric disease
* Pregnancy
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
Total Opioid Consumption in the First 24 Hours | 0-24 hours postoperatively
  The cumulative amount of opioid analgesic (fentanyl via patient-controlled analgesia device) used by each patient during the first 24 hours after laparoscopic cholecystectomy. This measure will evaluate the effectiveness of each intervention in reducing postoperative opioid requirement.

SECONDARY OUTCOMES:
Postoperative Pain Scores (Visual Analog Scale, VAS) | At 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24 hours postoperatively
  Pain intensity will be assessed using the Visual Analog Scale (VAS, 0-10 ; 0 = no pain, 10 = worst imaginable pain) during active (movement) and passive (rest) conditions.
Incidence of Postoperative Nausea and Vomiting (PONV) | 0-24 hours postoperatively
  Presence or absence of nausea and vomiting will be recorded to evaluate intervention-related side effects.
Incidence of Pruritus | 0-24 hours postoperatively
  Occurrence of itching will be recorded as a side effect possibly related to intrathecal morphine.
Incidence of Respiratory Depression | 0-24 hours postoperatively
  Respiratory depression will be defined as a respiratory rate < 8 breaths/min or oxygen saturation < 90% requiring intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Havva Yavuz Kayık, assistant doctor, Study Director — Ataturk University Department of Anesthesiology and Reanimation
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves sensitive patient health information, and data confidentiality will be strictly maintained according to institutional ethical guidelines.

REFERENCES:
- [Background] Motamed C, Bouaziz H, Franco D, Benhamou D. Analgesic effect of low-dose intrathecal morphine and bupivacaine in laparoscopic cholecystectomy. Anaesthesia. 2000 Feb;55(2):118-24. doi: 10.1046/j.1365-2044.2000.055002118.x. PMID 10651671
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Altuntas G, Akkaya OT, Ozkan D, Sayin MM, Balas S, Ozlu E. Comparison of Intraabdominal and Trocar Site Local Anaesthetic Infiltration on Postoperative Analgesia After Laparoscopic Cholecystectomy. Turk J Anaesthesiol Reanim. 2016 Dec;44(6):306-311. doi: 10.5152/TJAR.2016.75983. Epub 2016 Dec 1. PMID 28058142
- [Background] Ahmed SM, Shabbir S, Rana NA, Khatoon A, Ghani UF, Basharat I, Khan MN, Hameed FM, Dar MF. Ideal Local Anesthetic for Intraperitoneal Gallbladder Bed Infiltration Following Laparoscopic Cholecystectomy: A Randomized Controlled Trial. Cureus. 2024 Oct 9;16(10):e71122. doi: 10.7759/cureus.71122. eCollection 2024 Oct. PMID 39525126
- [Background] Kehlet H, Dahl JB. Anaesthesia, surgery, and challenges in postoperative recovery. Lancet. 2003 Dec 6;362(9399):1921-8. doi: 10.1016/S0140-6736(03)14966-5. PMID 14667752